CLINICAL TRIAL: NCT03622892
Title: Universal Haplotype-Based Non Invasive Prenatal Diagnosis by Linked-Read Sequencing (10XGenomics™ Technology)
Brief Title: Non-invasive Prenatal Diagnosis of Monogenic Disorders by Linked-reads Technology
Acronym: NID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: NID ( 29BRC18.0055)
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: Non Invasive Prenatal Diagnosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Parental DNA Maternal cell-free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Description of the presence of cell-free fetal DNA in maternal plasma allowed the possibility of non-invasive prenatal diagnosis. Whereas detection of paternally-inherited alleles is straightforward and being quickly implemented in routine, detection of maternally-inherited alleles remains challenging.

To date, the main approach that is being developped, called Relative Haplotype Dosage Analysis, relies on the identification of an allelic imbalance between the mother's wild-type and mutant alleles, relative to the fetal's contribution. This approach therefore requires the study of a propositus to identify the morbid haplotype, which is not always possible in the context of an ongoing pregnancy.

In this study, we aim to evaluate the contribution of new technologies, such as linked-read Sequencing, to allow direct identification of parental haplotype in the context of non-invasive prenatal diagnosis.

DETAILED DESCRIPTION:
Objectives:

The description of cell-free fetal DNA in maternal plasma offered the possibility of a non invasive approach for prenatal diagnosis (Non Invasive Prenatal Diagnosis, NIPD). However, only a small fraction of total cell-free DNA is of fetal origin, and its study widened only recently with the development of new technologies, such as digital PCR and Massively Parallel Sequencing.

Circulating fetal cells (CFC) represent a promising approach, but need further development before routine implementation To date, clinical applications are limited to Non Invasive Prenatal Testing for fetal aneuploidy and non invasive detection of fetal-specific genomic regions, for example fetal sex determination or fetal RHD genotyping, or more recently de novo mutations that can be suspected after echographic findings, such as achondroplasia. Yet, NIPD of maternally-inherited monogenic diseases remains challenging, for the fetal allele is hidden within a large amount of identical maternal sequences. Some publications report successful NIPD of maternally-inherited monogenic diseases, but only on case reports or small cohorts, without a standardized protocol and control of statistical risks.

In this study, we aim :

* to develop a new non invasive approach to Prenatal Diagnosis using both direct and indirect strategy by Massively Parallel Sequencing,
* to identify and characterize CFC.

Methods:

We recently acquired the Chromium™ technology (10XGenomics™). This approach, relying on microfluidic-based linked-read sequencing, allows direct haplotype phasing from long input DNA molecules, in this case parental genomic DNA. It is therefore possible to identify the mutant-linked haplotype for each parent and deduce fetal status with concomitant plasma DNA analysis.

We plan to include couples at risk of transmitting cystic fibrosis, during genetic counseling for prenatal diagnosis (PND). Non invasive analysis will be performed concomitantly to conventional PND, which will be performed on invasive fetal sample. After sequencing, we will use a new analysis algorithm that allows strict control of statistical risk.

Furthermore, we plan on using the Chromium Single Cell Solution (10XGenomics™) to isolate CFC. This approach allows analysis of single cell gene expression from thousands cells in a sample.

Expected results:

In this first study, we wish to include 20 couples in the course of 12 months, which will represent the largest cohort published to date.

We aim to assess feasibility of this new promising technology of Universal Haplotyping by linked-read sequencing in the context of NIPD of monogenic diseases, in terms of result accuracy as well as analysis time and technical cost. This straightforward protocol opens perspectives for a first-intention non invasive approach of prenatal diagnosis of familial monogenic diseases.

The Single Cell Solution will also enable us to differentiate the cell types circulating in maternal blood, and to identify molecular markers to isolate CFC.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies at 25% risk of being affected by Cystic Fibrosis with previously identified pathogenic variants
* Couple asking for invasive prenatal diagnosis
* Pregnancy at 8 weeks of gestation or later

Exclusion Criteria:

* Couple not asking for prenatal diagnosis
* No signed consent obtained

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Couples at 25% risk of transmitting Cystic Fibrosis and asking for prenatal diagnosis for this indication in the pluridisciplinary centers of Brest, Nantes, Dijon or Rouen University Hospitals, France.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-10-18 (Estimated); Study Completion 2021-10-18 (Estimated)

PRIMARY OUTCOMES:
Non-invasive Prenatal Diagnosis of Monogenic Disorders | 3 years
  Development of a robust and standardized NIPD protocol relying on Relative Haplotype Dosage Analysis after deciphering of parental haplotype by Linked-Read Sequencing

SECONDARY OUTCOMES:
Description of Circulating Fetal Cells | 3 years
  Use of the 10X Genomics* Single Cell Solution to identify Circulating Fetal Cells and describe their transcriptional characteristics in order to develop a cell-based Non Invasive Prenatal Diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Claude Ferec, MD, PhD, Study Director — CHU de Brest
Locations (6):
- France (6):
  - CHRU de Brest, Brest
  - CHRU de Dijon, Dijon
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CH Saint Brieuc, Saint-Brieuc